CLINICAL TRIAL: NCT04070170
Title: The Effects of Lower Level Laser Therapy on Orthodontic Tooth Movement
Brief Title: Laser Therapy on Orthodontic Tooth Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ildeu Andrade Jr. (Other)
Responsible Party: Sponsor-Investigator, Ildeu Andrade Jr., Professor, Pontifícia Universidade Católica de Minas Gerais
Organization: Pontifícia Universidade Católica de Minas Gerais (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Laser on tooth movement
Record Dates: First submitted 2019-08-15; First posted 2019-08-28 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Laser Therapy; Orthodontic Tooth Movement; Bone Remodeling
Keywords: Low-Level Light Therapy; Tooth Movement; Bone Remodeling
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (5):
- Low-level laser therapy and no orthodontic force (Experimental): No orthodontic force. Laser is applied on the first day and the premolars is extracted after 24 hours
  Interventions: Device: Low-level Laser Therapy
- Low-level laser therapy and application of orthodontic force (Experimental): Orthodontic force and Laser is applied on the first day and the premolars is extracted after 24 hours
  Interventions: Device: Low-level Laser Therapy; Procedure: Orthodontic force
- Orthodontic force only (Active Comparator): Orthodontic force is applied and the premolars is extracted after 24 hours, with no laser therapy
  Interventions: Procedure: Orthodontic force
- Low-level laser therapy and orthodontic force (Experimental): Orthodontic force and Laser is applied and the orthodontic tooth movement is evaluated
  Interventions: Device: Low-level Laser Therapy; Procedure: Orthodontic force
- Orthodontic force with no laser therapy (Active Comparator): Orthodontic force is applied and the orthodontic tooth movement is evaluated, with no laser therapy
  Interventions: Procedure: Orthodontic force

INTERVENTIONS:
Device: Low-level Laser Therapy — Low-level laser therapy is applied on premolars that will be extracted for treatment plan reasons
  Arms: Low-level laser therapy and application of orthodontic force; Low-level laser therapy and no orthodontic force; Low-level laser therapy and orthodontic force
Procedure: Orthodontic force — Mechanical loading is applied on premolars that will be extracted for treatment plan reasons and in canines for tooth movement
  Arms: Low-level laser therapy and application of orthodontic force; Low-level laser therapy and orthodontic force; Orthodontic force only; Orthodontic force with no laser therapy

SUMMARY:
The aims of this study will be to evaluate if a Lower Level Laser Therapy (LLLT): (1) enhances the levels of important pro-inflammatory chemokines involved in the bone remodeling process; (2) increases the rate of orthodontic tooth movement (OTM) on human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Facial convexity
* Protrusion or biprotrusion of the incisors
* Dental crowding
* Healthy periodontal condition
* Satisfactory oral hygiene

Exclusion Criteria:

* Patients under medications that may interfere with bone metabolism, such as anti-inflammatory, antibiotics and hormonal supplements in the previous three months
* Skeletal crossbite
* Parafunctional habits
* Occlusal interference

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2018-11-06 (Actual); Study Completion 2019-09-16 (Actual)

PRIMARY OUTCOMES:
Rate of orthodontic tooth movement, with and without low-level laser therapy | The quantification of OTM was performed before canine retraction
  The canine retraction was measured with a digital dynamometer
Rate of orthodontic tooth movement, with and without low-level laser therapy | The quantification of OTM was performed after 1 month of canine retraction
  The canine retraction was measured with a digital dynamometer
Rate of orthodontic tooth movement, with and without low-level laser therapy | The quantification of OTM was performed after 2 months of canine retraction
  The canine retraction was measured with a digital dynamometer
Rate of orthodontic tooth movement, with and without low-level laser therapy | The quantification of OTM was performed after 3 months of canine retraction
  The canine retraction was measured with a digital dynamometer

SECONDARY OUTCOMES:
Chemokine levels in the periodontal tissue after LLLT and orthodontic force | The chemokine levels were assayed on days 0, 1, 7 and 14 after application of orthodontic force and low-level laser therapy
  The chemokine levels were measured in the periodontal tissue after LLLT and orthodontic force by means of a cytometric bead array (CBA)

CONTACTS AND LOCATIONS:
Locations (1):
- Pontifical Catholic University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doshi-Mehta G, Bhad-Patil WA. Efficacy of low-intensity laser therapy in reducing treatment time and orthodontic pain: a clinical investigation. Am J Orthod Dentofacial Orthop. 2012 Mar;141(3):289-297. doi: 10.1016/j.ajodo.2011.09.009. PMID 22381489
- [Background] Alhashimi N, Frithiof L, Brudvik P, Bakhiet M. Chemokines are upregulated during orthodontic tooth movement. J Interferon Cytokine Res. 1999 Sep;19(9):1047-52. doi: 10.1089/107999099313271. PMID 10505748
- [Background] Torri S, Weber JB. Influence of low-level laser therapy on the rate of orthodontic movement: a literature review. Photomed Laser Surg. 2013 Sep;31(9):411-21. doi: 10.1089/pho.2013.3497. Epub 2013 Jul 24. PMID 23883115
- [Background] Genc G, Kocadereli I, Tasar F, Kilinc K, El S, Sarkarati B. Effect of low-level laser therapy (LLLT) on orthodontic tooth movement. Lasers Med Sci. 2013 Jan;28(1):41-7. doi: 10.1007/s10103-012-1059-6. Epub 2012 Feb 18. PMID 22350425
- [Background] Kim SJ, Moon SU, Kang SG, Park YG. Effects of low-level laser therapy after Corticision on tooth movement and paradental remodeling. Lasers Surg Med. 2009 Sep;41(7):524-33. doi: 10.1002/lsm.20792. PMID 19639625